CLINICAL TRIAL: NCT04051554
Title: Effect of Neuromuscular and Proprioceptive Training in Reducing Landing Error Patterns in Football Players
Brief Title: Neuromuscular and Proprioceptive Training in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RiphahIU Hafiz Ali Bin Asim
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Football Players; Sport Injury; Sports Physical Therapy
Keywords: ACL Injury; Landing Error Score System; Neuromuscular Training; Proprioceptive Training; Soccer
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular and Proprioceptive Training (Experimental): Myklebust's training program
  Interventions: Other: Neuromuscular and Proprioceptive Training
- Conventional Training (Active Comparator): Running, Sprints, Agility training, and Dynamic stretching
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Neuromuscular and Proprioceptive Training — Myklebust's training program (floor exercises, mat exercises, and wobble board exercises for 5 weeks)
  Arms: Neuromuscular and Proprioceptive Training
Other: Conventional Training — Running, Sprinting, Agility training and Dynamic stretching for five weeks
  Arms: Conventional Training

SUMMARY:
The objective of this study was to determine the effect of proprioceptive and neuromuscular training on landing errors and balance of the football players. This was randomized controlled trial in which 40 football players were randomly allocated into experimental and control group. The control group followed conventional exercise plan while experimental group players were being trained under Myklebust's training program. Data were collected at baseline and after follow-up of five weeks Landing Error Score System (LESS) and Biodex Single Leg Stability (SLS) score. Data were analyzed using statistical package for social sciences (SPSS)-21.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injuries are a severe public health issue from both an economic and general wellness view. This burden will be reduced by promoting compliance and the use of injury prevention programs. To reduce injury rates, trainers, athletes, parents, and the team of sports medicine need to know the advantages of injury prevention programs. Parents and employees in sports medicine want a program that can decrease the risk of injury. Coaches and athletes are looking for a program that will also increase athletic efficiency without taking time off exercise, time that would otherwise be spent honing sport-specific abilities. Injury prevention programs in youth athletics will promote neuromuscular enhancements and create appropriate long-term techniques while instantly preparing the athlete for competition.

Various studies have been done to assess the role of proprioceptive and neuromuscular exercises on reducing incidence of ACL injury. No conclusive result has been established as yet that these type of exercises really reduce the incidence of ACL injury or not. However, it is found that by performing certain exercises there is improvement in biomechanics of jump landing as predicted by LESS score which is a reliable tool to establish risk of ACL and other lower limb injury in an athlete. Therefore the investigators have used a lower limb injury prevention program to assess its effectiveness in reducing LESS score.

ELIGIBILITY:
Inclusion Criteria:

* Male football players registered with Pakistan Sports Board, Islamabad.
* Players playing for a minimum of 20 hrs per week.
* The participant should understand and sign the informed consent form.
* Players should agree to take part in the training program for 35 days.

Exclusion Criteria:

* Players with any major neuromusculoskeletal or cardiovascular pathology in last 6 months.
* Players having any psychological issue

Ages: 15 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Unavailability of the female athletes in our setting
Enrollment: 40 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Landing Error Score System (LESS) | 5th week
  Changes for the baseline, there are 17 items in LESS. Maximum possible score is 19 which show very poor mechanics and score of 5 and less than 5 are considered good to excellent.
Single Leg Stability | 5th week
  Measures were obtained from 20-sec trials during which participants were asked to maintain an upright standing position on their dominant limb on the unstable surface of the Biodex Stability and Balance System.Its reliability is R = .94

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, DSc (PT), Principal Investigator — Riphah International university, Islamabad
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franklin CC, Weiss JM. Stopping sports injuries in kids: an overview of the last year in publications. Curr Opin Pediatr. 2012 Feb;24(1):64-7. doi: 10.1097/MOP.0b013e32834ec618. PMID 22227777
- [Background] Injuries in youth soccer: a subject review. American Academy of Pediatrics. Committee on Sports Medicine and Fitness. Pediatrics. 2000 Mar;105(3 Pt 1):659-61. PMID 10699129
- [Background] Nettle H, Sprogis E. Pediatric exercise: truth and/or consequences. Sports Med Arthrosc Rev. 2011 Mar;19(1):75-80. doi: 10.1097/JSA.0b013e318209cf2b. PMID 21293241
- [Background] Schub D, Saluan P. Anterior cruciate ligament injuries in the young athlete: evaluation and treatment. Sports Med Arthrosc Rev. 2011 Mar;19(1):34-43. doi: 10.1097/JSA.0b013e31820b960d. PMID 21293236
- [Background] Hill DE, Andrews JR. Stopping sports injuries in young athletes. Clin Sports Med. 2011 Oct;30(4):841-9. doi: 10.1016/j.csm.2011.07.003. No abstract available. PMID 22018324
- [Background] DiFiori JP. Evaluation of overuse injuries in children and adolescents. Curr Sports Med Rep. 2010 Nov-Dec;9(6):372-8. doi: 10.1249/JSR.0b013e3181fdba58. PMID 21068572
- [Background] Leininger RE, Knox CL, Comstock RD. Epidemiology of 1.6 million pediatric soccer-related injuries presenting to US emergency departments from 1990 to 2003. Am J Sports Med. 2007 Feb;35(2):288-93. doi: 10.1177/0363546506294060. Epub 2006 Nov 7. PMID 17092927
- [Background] Knowles SB, Marshall SW, Miller T, Spicer R, Bowling JM, Loomis D, Millikan RW, Yang J, Mueller FO. Cost of injuries from a prospective cohort study of North Carolina high school athletes. Inj Prev. 2007 Dec;13(6):416-21. doi: 10.1136/ip.2006.014720. PMID 18056320
- [Background] Hewett TE, Ford KR, Hoogenboom BJ, Myer GD. Understanding and preventing acl injuries: current biomechanical and epidemiologic considerations - update 2010. N Am J Sports Phys Ther. 2010 Dec;5(4):234-51. PMID 21655382
- [Background] Carter CW, Micheli LJ. Training the child athlete: physical fitness, health and injury. Br J Sports Med. 2011 Sep;45(11):880-5. doi: 10.1136/bjsports-2011-090201. PMID 21836172